CLINICAL TRIAL: NCT05703750
Title: Impact of Clinical Evident Portal Hypertension on Hepatocellular Carcinoma With Transarterial Chemoembolization (CHANCE-CHESS 2301): A Multicenter Retrospective Study
Brief Title: Impact of Clinical Evident Portal Hypertension on HCC With TACE (CHANCE-CHESS 2301)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE-CHESS 2301
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma; Portal Hypertension
Keywords: hepatocellular carcinoma; transarterial chemoembolization; clinical evident portal hypertension
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEPH group: CEPH was defined when at least one following factor was present: 1) esophageal/gastric varices on upper endoscopy or CT imaging, 2) ascites requiring diuretic treatment, 3) splenomegaly (largest diameter on CT >12 cm) with a low platelet count (<100,000/mm3).
  Interventions: Procedure: TACE ± Systemic therapy
- non-CEPH group: Non-CEPH was defined when none of the following factor was present: 1) esophageal/gastric varices on upper endoscopy or CT imaging, 2) ascites requiring diuretic treatment, 3) splenomegaly (largest diameter on CT >12 cm) with a low platelet count (<100,000/mm3).
  Interventions: Procedure: TACE ± Systemic therapy

INTERVENTIONS:
Procedure: TACE ± Systemic therapy — TACE: cTACE (conventional TACE) or dTACE (drug-eluting beads TACE); Systemic therapy: PD-1/PD-L1 inhibitors, VEGF-TKI/bevacizumab, PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab, radiotherapy or chemotherapy.

SUMMARY:
The purpose of this study is to discuss the prognostic value of CEPH among HCC patients underwent TACE treatment, its impact on overall survival, and try to stratify patient cohorts for a better treatment strategy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer worldwide and the second leading cause of cancer-related deaths globally. Transarterial chemoembolization (TACE) is recommended as standard therapy for intermediate-stage HCC according to the current guidelines and is also the most widely used in advanced HCC in real-world practice. Clinically relevant portal hypertension increases the risk of hepatic decompensation, which impairs survival in patients with HCC. The purpose of this study is to discuss the prognostic value of CEPH among HCC patients who underwent TACE treatment, its impact on overall survival, and try to stratify patient cohorts for a better treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Received at least 1 TACE treatment；

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. ECOG Performance Score > 2;
3. History of spleen resection;
4. Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC treated with TACE ± Systemic Treatment from June 2006 to December 2021.
Sampling Method: Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any treatment to death due to any cause.

SECONDARY OUTCOMES:
Objective response rate(ORR) per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per mRECIST.
Progression free survival(PFS) per mRECIST | up to approximately 2 years
  The PFS is defined as the time from the initiation of any treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China; Xiaolong Qi, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (2):
- China (2):
  - Gao-Jun Teng, Nanjing
  - Xiaolong Qi, Nanjing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez-Gea V, Turon F, Berzigotti A, Villanueva A. Management of small hepatocellular carcinoma in cirrhosis: focus on portal hypertension. World J Gastroenterol. 2013 Feb 28;19(8):1193-9. doi: 10.3748/wjg.v19.i8.1193. PMID 23482437
- [Background] Muller L, Hahn F, Mahringer-Kunz A, Stoehr F, Gairing SJ, Foerster F, Weinmann A, Galle PR, Mittler J, Pinto Dos Santos D, Pitton MB, Duber C, Fehrenbach U, Auer TA, Gebauer B, Kloeckner R. Prevalence and clinical significance of clinically evident portal hypertension in patients with hepatocellular carcinoma undergoing transarterial chemoembolization. United European Gastroenterol J. 2022 Feb;10(1):41-53. doi: 10.1002/ueg2.12188. Epub 2021 Dec 16. PMID 34918471
- [Background] Faitot F, Allard MA, Pittau G, Ciacio O, Adam R, Castaing D, Cunha AS, Pelletier G, Cherqui D, Samuel D, Vibert E. Impact of clinically evident portal hypertension on the course of hepatocellular carcinoma in patients listed for liver transplantation. Hepatology. 2015 Jul;62(1):179-87. doi: 10.1002/hep.27864. Epub 2015 May 20. PMID 25914217
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438